CLINICAL TRIAL: NCT05585632
Title: Phase 1, Randomized, Observer-blind Study to Evaluate the Safety, Reactogenicity, and Immunogenicity of Multi-component Vaccines mRNA-1045 (Influenza and RSV) or mRNA-1230 (Influenza, RSV, and SARS-CoV-2) Compared With mRNA-1010 (Influenza), mRNA-1345 (RSV), and mRNA-1273.214 (SARS-CoV-2) Vaccines in Healthy Adults 50-75 Years of Age
Brief Title: A Safety, Reactogenicity, and Immunogenicity Study of mRNA-1045 (Influenza and Respiratory Syncytial Virus [RSV]) or mRNA-1230 (Influenza, RSV, and Severe Acute Respiratory Syndrome Coronavirus 2 [SARS-CoV-2]) Vaccine in Adults 50 to 75 Years Old
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ModernaTX, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: mRNA-1230-P101; 2022-002138-15 (EudraCT Number)
Record Dates: First submitted 2022-10-14; First posted 2022-10-19 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2024-03

CONDITIONS: SARS-CoV-2; Influenza; RSV
Keywords: mRNA-1230 Vaccine; mRNA-1045 Vaccine; SARS-CoV-2 Vaccine; Influenza Vaccine; RSV Vaccine; Coronavirus; Virus Diseases; Messenger RNA; COVID-19; COVID-19 Vaccine; Moderna
MeSH Terms: conditions — Influenza, Human; Coronavirus Infections; Virus Diseases; COVID-19 | interventions — mRNA-1010 influenza vaccine; mRNA-1345 respiratory syncytial virus vaccine; mRNA-1273.214 COVID-19 vaccine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: All participants will be unblinded at Day 29 (1 month following study injection) to seek immunization with licensed influenza and/or SARS-CoV-2 vaccines, outside of the study, per local standard of care.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (9):
- mRNA-1010 (Experimental): Participants will receive a dose of mRNA-1010 by intramuscular (IM) injection on Day 1.
  Interventions: Biological: mRNA-1010
- mRNA-1345 (Experimental): Participants will receive a dose of mRNA-1345 by IM injection on Day 1.
  Interventions: Biological: mRNA-1345
- mRNA-1273.214 (Experimental): Participants will receive a dose of mRNA-1273.214 by IM injection on Day 1.
  Interventions: Biological: mRNA-1273.214
- mRNA-1045 Dose Level A (Experimental): Participants will receive mRNA-1045 at Dose Level A by IM injection on Day 1.
  Interventions: Biological: mRNA-1045
- mRNA-1045 Dose Level B (Experimental): Participants will receive mRNA-1045 at Dose Level B by IM injection on Day 1.
  Interventions: Biological: mRNA-1045
- mRNA-1045 Dose Level C (Experimental): Participants will receive mRNA-1045 at Dose Level C by IM injection on Day 1.
  Interventions: Biological: mRNA-1045
- mRNA-1230 Dose Level A (Experimental): Participants will receive mRNA-1230 at Dose Level A by IM injection on Day 1.
  Interventions: Biological: mRNA-1230
- mRNA-1230 Dose Level B (Experimental): Participants will receive mRNA-1230 at Dose Level B by IM injection on Day 1.
  Interventions: Biological: mRNA-1230
- mRNA-1230 Dose Level C (Experimental): Participants will receive mRNA-1230 at Dose Level C by IM injection on Day 1.
  Interventions: Biological: mRNA-1230

INTERVENTIONS:
Biological: mRNA-1010 — Sterile liquid for injection
  Arms: mRNA-1010
Biological: mRNA-1345 — Sterile liquid for injection
  Arms: mRNA-1345
Biological: mRNA-1273.214 — Sterile liquid for injection
  Arms: mRNA-1273.214
Biological: mRNA-1045 — Formulation for injection
  Arms: mRNA-1045 Dose Level A; mRNA-1045 Dose Level B; mRNA-1045 Dose Level C
Biological: mRNA-1230 — Formulation for injection
  Arms: mRNA-1230 Dose Level A; mRNA-1230 Dose Level B; mRNA-1230 Dose Level C

SUMMARY:
The primary goal of this study is to evaluate the safety and reactogenicity of multi-component vaccines mRNA-1045 (Influenza and RSV) and mRNA-1230 (influenza, RSV, and SARS-CoV-2) compared with mRNA-1010 (influenza), mRNA-1345 (RSV), and mRNA-1273.214 (SARS-CoV-2) vaccines in healthy older participants.

ELIGIBILITY:
Inclusion Criteria:

* Investigator assessment that participant understands and is willing and physically able to comply with protocol-mandated follow-up, including all procedures.
* Body mass index of 18 to 35 kilograms/square meter (kg/m^2) (inclusive) at the Screening Visit(s).
* For female participants of childbearing potential: negative pregnancy test, adequate contraception or has abstained from all activities that could result in pregnancy for at least 28 days prior to Day 1, agreement to continue adequate contraception or abstinence through 3 months following the vaccination, and not currently breastfeeding.
* Fully vaccinated for COVID-19 with an approved primary series according to the locally authorized or approved regimen. The most recent COVID-19 vaccine (primary series or booster) must be ≥120 days before (or less per local guidance) Day 1.

Exclusion Criteria:

* Acutely ill or febrile (temperature ≥38.0°Celsius/[100.4°Fahrenheit]) 72 hours before or at the Screening Visit or Day 1. Participants meeting this criterion may be rescheduled within the 28-day screening window for re-evaluation and will retain their initially assigned participant number.
* Any medical, psychiatric, or occupational condition, including reported history of drug or alcohol abuse, that, in the opinion of the investigator, might pose additional risk due to participation in the study or could interfere with the interpretation of study results.
* Has received systemic immunosuppressants or immune-modifying drugs for >14 days in total within 6 months before screening (for corticosteroids ≥10 milligrams (mg)/day of prednisone or equivalent) or is anticipating the need for immunosuppressive treatment at any time during participation in the study.
* Received or plans to receive any vaccine authorized or approved by a local health agency ≤28 days before study injections (Day 1) or within 28 days after the study injection.
* Received a licensed seasonal influenza vaccine or any other investigational influenza or RSV vaccine within ≤180 days before Day 1.
* Tested positive for influenza or RSV by local health authority-approved testing methods within ≤180 days before Day 1.
* Significant exposure to someone with SARS-CoV-2 infection or COVID-19 in the past 14 days, as defined by the United States Center for Disease Control (CDC) or the European Centre for Disease Prevention and Control as a high risk (close contact) of a COVID-19 case or known history of SARS-CoV-2 infection within the past 90 days before Day 1.
* Donated ≥450 mL of blood products within 28 days before the Screening Visit or plans to donate blood products during the study.

Note: Other inclusion and exclusion criteria may apply.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 392 (Actual)
Dates: Start 2022-10-14 (Actual); Primary Completion 2024-02-28 (Actual); Study Completion 2024-02-28 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Solicited Local and Systemic Adverse Reactions (ARs) | Up to Day 8 (7 days post vaccination)
Number of Participants with Unsolicited Adverse Events (AEs) | Up to Day 29 (28 days post vaccination)
Number of Participants with Medically-Attended AEs (MAAEs) | Day 1 through Day 361
Number of Participants with Adverse Events of Special Interest (AESIs) | Day 1 through Day 361
Number of Participants with Serious Adverse Events (SAEs) | Day 1 through Day 361
Number of Participants with AEs Leading to Discontinuation | Day 1 through Day 361

SECONDARY OUTCOMES:
Change From Baseline in Geometric Mean Titer (GMT) as Measured by Hemagglutination Inhibition (HAI) Assay at Day 29 | Baseline (Day 1), Day 29
Change From Baseline in GMT as Measured by Pseudovirus Neutralization Assay (PsVNA) (or Binding Antibody Assay) at Day 29 | Baseline (Day 1), Day 29
Change From Baseline in GMT as Measured by Microneutralization Assay at Day 29 | Baseline (Day 1), Day 29
Change From Baseline in Geometric Mean Fold-Rise (GMFR) as Measured by HAI Assay at Day 29 | Baseline (Day 1), Day 29
Change From Baseline in GMFR as Measured by PsVNA (or Binding Antibody Assay) at Day 29 | Baseline (Day 1), Day 29
Change From Baseline in GMFR as Measured by Microneutralization Assay at Day 29 | Baseline (Day 1), Day 29
Influenza: Percentage of Participants with Seroconversion as Measured by HAI Assay | Baseline (Day 1) to Day 29
  Seroconversion is defined as a Day 29 titer ≥1:40 if baseline is <1:10 or a 4-fold or greater rise if baseline is ≥1:10 in anti-HA antibodies measured by HAI assay.
SARS-CoV-2: Percentage of Participants with Seroresponse as Measured by PsVNA (or Binding Antibody Assay) | Baseline (Day 1) to Day 29
  Seroresponse is defined as a Day 29 titer ≥4-fold if baseline is ≥lower limit of quantification (LLOQ) or ≥4*LLOQ if baseline titer is <LLOQ in nAb titers measured by PsVNA (or binding antibody assay).
RSV: Percentage of Participants with Seroresponse as Measured by RSV Neutralization Assay | Baseline (Day 1) to Day 29
  Seroresponse is defined as a Day 29 titer ≥4-fold if baseline is ≥LLOQ or ≥4*LLOQ if baseline titer is <LLOQ in nAb titers measured by RSV neutralization assay.

CONTACTS AND LOCATIONS:
Locations (30):
- United States (14):
  - Accel Research Sites, DeLand, Florida
  - Research Centers of America (cenexel), Hollywood, Florida
  - Accel Research Sites, St. Petersburg, Florida
  - Atlanta Center for Medical Research - Family Medicine, Atlanta, Georgia
  - Centricity Research, Columbus, Georgia
  - Cenexel IRA (iResearch Atlanta), Decatur, Georgia
  - Optimal Research, Peoria, Illinois
  - DM Clinical Research, Southfield, Michigan
  - Lucas Research, Inc. (Diabetes & Endocrinology Consultants PC), Morehead City, North Carolina
  - Trial Management Associates, Wilmington, North Carolina
  - Velocity Clinical Research, Anderson, South Carolina
  - Trial Management Associates, Myrtle Beach, South Carolina
  - DM Clinical Research, Houston, Texas
  - DM Clinical Research, Sugar Land, Texas
- Australia (7):
  - Paratus Clinical Research Western Sydney, Blacktown, New South Wales
  - Paratus Clinical Kanwal, Kanwal, New South Wales
  - Paratus Clinical Research Brisbane, Albion, Queensland
  - Nucleus Network Brisbane Clinic - Centre For Clinical Studies, Herston, Queensland
  - University of the Sunshine Coast, South Brisbane, Queensland
  - AusTrials Taringa, Taringa, Queensland
  - Emeritus Research, Camberwell, Victoria
- United Kingdom (9):
  - Newcastle University - Institute of Cellular Medicine (ICM), Newcastle, England
  - Nottingham University Hospitals NHS Trust - Queen's Medical Centre (QMC) Campus, Nottingham, Nottinghamshire
  - University of Oxford, Oxford, Oxfordshire
  - Bristol Royal Hospital for Children, Bristol
  - Royal Devon & Exeter Hospital, Exeter
  - Chelsea and Westminster Hospital, London
  - St George's Healthcare NHS Trust - University of London - Th, London
  - National Hospital for Neurology and Neurosurgery, London
  - Southampton General Hospital, Southampton